CLINICAL TRIAL: NCT04606576
Title: A Double-Blinded, Placebo-controlled, Double Dummy, Multi-center Randomized, Phase 3 Study to Evaluate the Efficacy and Safety of ORMD-0801 in Subjects With T2DM With Inadequate Glycemic Control on 1, 2 or 3 Oral Glucose-lowering Agents.
Brief Title: Study to Evaluate the Efficacy and Safety of ORMD-0801 in Subjects With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: ORA-D-013-1 was terminated based on the primary results analyzed at the end of the treatment, week 26.
Sponsor: Oramed, Ltd. (Industry)
Collaborators: Integrium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORA-D-013-1
Record Dates: First submitted 2020-10-22; First posted 2020-10-28 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Fish Oils; Insulin

STUDY DESIGN:
Intervention Model Description: In this randomized, double-blind, double dummy, placebo-controlled study, approximately 675 eligible subjects with type 2 diabetes and inadequate control on at least one and up to 3 oral glucose-lowering agents will undergo an initial 21-day Screening Period, followed by a 26-week Double-Blind Treatment Period and a 26-week Double-Blind Treatment Extension Period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Fish Oil
  Interventions: Other: Placebo
- ORMD-0801 QD (Experimental): 8 mg ORMD-0801 administered QD at night
  Interventions: Drug: ORMD-0801 QD
- ORMD-0801 BID (Experimental): 8 mg ORMD-0801 administered at night and in the morning 45 minutes before breakfast.
  Interventions: Drug: ORMD-0801 BD

INTERVENTIONS:
Other: Placebo — Fish Oil
  Other Names: Fish Oil
  Arms: Placebo
Drug: ORMD-0801 QD — Oral Insulin once per day
  Other Names: Oral Insulin
  Arms: ORMD-0801 QD
Drug: ORMD-0801 BD — Oral Insulin, twice per day
  Other Names: Oral Insulin
  Arms: ORMD-0801 BID

SUMMARY:
In this randomized, double-blind, double-dummy, placebo-controlled study, approximately 675 eligible subjects with type 2 diabetes and inadequate control on at least one and up to 3 oral glucose-lowering agents will undergo an initial 21-day Screening Period, followed by a 26-week Double-Blind Treatment Period and a 26-week Double-Blind Treatment Extension Period.

DETAILED DESCRIPTION:
Screening Period Subjects will provide a written informed consent during Screening Visit 1. They will be scheduled to return to the clinic 10 days prior to randomization for Screening Visit 2. At this visit, a CGM sensor will be placed with appropriate instructions by the study team for a 10-day blinded CGM data collection by the site. Subjects will then return to the clinic after 10 days (± 1-day) for removal of the CGM sensor. The subjects will be randomized to one of the three arms of the study treatment.

3.1.2 26-Week Double-Blind Treatment Period After the Screening Period, subjects will be randomized to 26 weeks of the Double-Blind Treatment Period. In a double-blind, double dummy randomization scheme, subjects will either receive ORMD-0801 administered once-daily at night (1 x 8 mg capsule between 8 PM to 12 Midnight and no sooner than 1 hour after dinner); or ORMD-0801 8 mg (1 x 8 mg capsule) administered twice daily, each morning approximately 45 minutes (±15 minutes) prior to breakfast and each night prior to bedtime (between 8 PM to 12 Midnight and no sooner than 1 hour after dinner) or matching placebo. Subjects will receive 1 capsule approximately 45 minutes (±15 minutes) prior to breakfast and 1 capsule between 8 PM to 12 Midnight and no sooner than 1 hour after dinner.

During the Double-Blind Treatment Period commencing at Week 0 (Visit 1, CGM removal), subjects will return to the clinic at the following intervals: Week 6 - Visit 2; Week 12 - Visit 3; Week 18 -Visit 4; Week 24 - Visit 5 (10 days (± 1-day) prior to Week 26 for CGM application) and Week 26 - Visit 6 (CGM removal and end of Double-Blind Treatment Period visit).

The visit requiring CGM application will occur 10 days prior to the CGM removal visit within ± 1-day window.

3.1.3 26-Week Double-Blind Treatment Extension Period Following the completion of the Double-Blind Treatment Period, subject will enter a 26-week Double-Blind Treatment Extension Period. Subjects previously randomized to placebo during the Double-Blind Treatment Period will be randomized to receive either ORMD-0801 8 mg QD or 8 mg BID for the duration of the Double-Blind Treatment Extension Period. Subjects previously randomized to 8 mg QD or 8 mg BID during the Double-Blind Treatment Period will remain in the same treatment arm for the duration of the Double-Blind Treatment Extension Period. The Extension Period treatment assignments will remain blinded for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 - 75 years.
* Established diagnosis of T2DM for at least 6 months prior to Screening AND an A1C ≥ 7.5% but ≤ 11.0% at Screening.
* On a stable dose of at least one and up to three of the following oral glucose-lowering agents: Metformin, DPP-4 inhibitor, SGLT-2 inhibitor, thiazolidinedione, or sulfonylurea for a period of 3 months prior to Screening.
* Body mass index (BMI) of 25-40 kg/m2 at Screening and stable weight, with no more than 5 kg gain or loss in the 3 months prior to Screening.
* Renal function - GFR ≥ 30 ml/min/1.73 m2.
* Females of childbearing potential must:

  * a. have a negative serum pregnancy test result at Screening.
  * b. agree to avoid becoming pregnant while receiving IP for at least 30 days prior to IP administration, during the entire study, and for 30 days following their last dose of IP.
  * c. agree to use an acceptable method of contraception at least 30 days prior to IP administration, during the entire study, and for 30 days following their last dose of IP. Acceptable methods of contraception are hormonal contraception (contraceptive pill or injection) PLUS an additional barrier method of contraception such as a diaphragm, condom, sponge, or spermicide.
  * d. In the absence of hormonal contraception, double-barrier methods must be used which include a combination of any two of the following: diaphragm, condom, copper intrauterine device, sponge, or spermicide, and must be used for at least 30 days prior to administration of IP, during the entire study, and for 30 days following their last dose of IP.
  * e. Abstinence (relative to heterosexual activity) can be used as the sole method of contraception if it is consistently employed as the subject's preferred and usual lifestyle and if considered acceptable by local regulatory agencies and ERCs/IRBs. Periodic abstinence (e.g., calendar, ovulation, sympto-thermal, post-ovulation methods, etc.) and withdrawal are not acceptable methods of contraception.
  * f. Females who are not of childbearing potential are defined as:

    * i. Postmenopausal (defined as at least 12 months with no menses in women ≥45 years of age); OR
    * ii. Have had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal ligation/occlusion at least 6 weeks prior to screening; OR
    * iii. Have a congenital or acquired condition that prevents childbearing.

Exclusion Criteria:

Subjects with:

* Type 1 diabetes.
* A history of diabetes mellitus with ketoacidosis or is assessed by the Investigator as possibly having type 1 diabetes mellitus confirmed by a C-peptide < 0.4 ng/mL (0.13 nmol/L) at Screening.
* Diabetes attributable to other secondary causes (e.g., genetic syndromes, secondary pancreatic diabetes, diabetes due to endocrinopathies, drug- or chemical-induced, and post-organ transplant).
* Treatment involving glucosidase inhibitor, insulin secretagogues (other than sulfonylureas), or GLP-1 receptor agonists within 3 months prior to Visit 1.
* A history of >2 episodes of severe hypoglycemia within 6 months prior to Screening.
* A history of hypoglycemic unawareness.
* A history of unstable angina or myocardial infarction within 6 months prior to Screening, New York Heart Association (NYHA) Grade 3 or 4 congestive heart failure (CHF), valvular heart disease, ventricular cardiac arrhythmia requiring treatment, pulmonary hypertension, cardiac surgery, coronary angioplasty, stroke or transient ischemic attack (TIA) within 6 months prior to Screening.
* A history of uncontrolled or untreated severe hypertension defined as systolic blood pressure above or equal to 160 mmHg and/or diastolic blood pressure above or equal to 100 mmHg. A single repeat measurement will be permitted.
* Renal dysfunction: GFR < 30 mL/min/1.73 m2.
* Active proliferative retinopathy requiring treatment.
* Psychiatric disorders that, per Investigator judgment, may have impact on the safety of the subject or interfere with the subject's participation or compliance in the study.
* Laboratory abnormalities at Screening including:

  * a. C-peptide < 0.4 ng/mL.
  * b. Abnormal serum thyrotropin (TSH) levels below the lower limit of normal or >1.5X the upper limit of normal; a single repeat test is allowable.
  * c. Elevated liver enzymes (alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP)) >3X the upper limit of normal; a single repeat test is allowable.
  * d. Very high fasting triglyceride levels (>600 mg/dL); a single repeat test is allowable.
  * e. Any relevant abnormality that would interfere with the efficacy or the safety assessments during study treatment administration.
* Positive history of active liver disease (other than non-alcoholic hepatic steatosis), primary biliary cirrhosis, or active symptomatic gallbladder disease.
* Positive results for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C virus ribonucleic acid (RNA).
* Patient has active or history of neoplastic disease (except for adequately treated non-invasive basal cell and/or squamous cell carcinoma or carcinoma in situ of the cervix) within the past 5 years prior to Baseline.
* Use of the following medications:

  * a. History of use of any injectable or inhaled, basal, pre-mixed or prandial insulin (greater than 7 days) within 6 months prior to Screening.
  * b. Administration of thyroid preparations or thyroxine (except in subjects on stable replacement therapy) within 6 weeks prior to Screening.
  * c. Requirements (in the last 12 months), or may require, systemic (oral, intravenous, intramuscular) glucocorticoid therapy for more than 2 weeks during the study period. Intra-articular and/or topical corticosteroids are not considered systemic.
  * d. Use of medications known to modify glucose metabolism or to decrease the ability to recover from hypoglycemia such as oral, parenteral, and immunosuppressive or immunomodulating agents. Inhaled nasal steroids are permissible.
* Known allergy to soy.
* Involvement in a weight loss program and is not in the maintenance phase, or subject has started weight loss medication (e.g., orlistat or liraglutide) within 3 months prior to Screening.
* Prior bariatric surgery.
* Subject is pregnant or breast-feeding.
* Subject is a user of recreational or illicit drugs or has had a recent history (within 1 year of Screening) of drug or alcohol abuse or dependence. (Note: Alcohol abuse includes heavy alcohol intake as defined by >3 drinks per day or >14 drinks per week or binge drinking) at Screening. Occasional intermittent use of cannabinoid products will be allowed provided that no cannabinoid products have been used during the 1 week prior to each visit.
* Contraindications to metformin use as per label.
* A history of gastrointestinal disorders (e.g. hypochlorhydria) with the potential to interfere with drug absorption.
* Any condition or other factor (at the Investigator's discretion) that is deemed unsuitable for subject enrollment into the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 710 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in A1C | Baseline and 26 Weeks
  The mean change from baseline (Visit 1) in A1C at 26 weeks (Visit 6) for the active and placebo groups.

SECONDARY OUTCOMES:
Mean change in fasting glucose | Baseline and 26 weeks
  The Mean change from baseline (Visit 1) in fasting plasma glucose at 26 weeks (Visit 6) will be analyzed using a linear mixed model similar to the primary analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Kidron, PhD, Study Director — Oramed, Ltd.
Locations (1):
- Orange County Research Center (OCRC) 14351 Myford Rd., Suite B, Tustin, CA 92780, Tustin, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2020. Diabetes Care. 2020 Jan;43(Suppl 1):S14-S31. doi: 10.2337/dc20-S002. PMID 31862745
- [Background] Cleary PA, Orchard TJ, Genuth S, Wong ND, Detrano R, Backlund JY, Zinman B, Jacobson A, Sun W, Lachin JM, Nathan DM; DCCT/EDIC Research Group. The effect of intensive glycemic treatment on coronary artery calcification in type 1 diabetic participants of the Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Study. Diabetes. 2006 Dec;55(12):3556-65. doi: 10.2337/db06-0653. PMID 17130504
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Nathan DM, Buse JB, Davidson MB, Heine RJ, Holman RR, Sherwin R, Zinman B. Management of hyperglycemia in type 2 diabetes: A consensus algorithm for the initiation and adjustment of therapy: a consensus statement from the American Diabetes Association and the European Association for the Study of Diabetes. Diabetes Care. 2006 Aug;29(8):1963-72. doi: 10.2337/dc06-9912. No abstract available. PMID 16873813